CLINICAL TRIAL: NCT06708546
Title: Study the Efficiency of Oral Nutritional Supplementation on Nutrition Status, Digestive Disorders, Respiratory Infection and Anorexic in Children Between 24 - 59 Months Old.
Brief Title: Improvement of Nutrition, Digestion, and Respiration in Children in Vietnam Using Oral Nutritional Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tu Nguyen Song (Other Government)
Responsible Party: Sponsor-Investigator, Tu Nguyen Song, Head of Division Planning, National Institute of Nutrition, Vietnam
Organization: National Institute of Nutrition, Vietnam (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: DIELACGROW-NIN
Record Dates: First submitted 2023-07-05; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Undernutrition; Wasting; Malnourished
Keywords: Picky eating; Children; Digestive condition; Respiratory condition; Wasting; Nutrient status
MeSH Terms: conditions — Malnutrition; Cachexia; Food Fussiness

STUDY DESIGN:
Intervention Model Description: Step 1: Investigate the nutritional status of all children aged 24 - 59 months in 6 selected communes in Yen Bai province. Expecting 2000 participants in 6 examined communes.
  Step 2: After the investigative selection, participants that meet the standard will be invited to the study ( the selected communes can be narrowed if the targets are met). The study will move to the next step when parents sign the consent paper.
  Step 3: Groups will be divided to investigate activities. Creating a list for all participants that meet the criteria, with Z-score height for age <-1 and Z-score weight for height<1. Random selection based on age ensures no significant difference in the nutritional index or related indicators in the group to assess the effectiveness of the intervention (divided by class/age). Then, randomly divided the target by class into two large groups (500 targets per group)
Who Masked: Participant, Investigator
Masking Description: Control Group (490 participants): children eating normally (not using Oral Nutritional Supplementation) during 4 months of intervention. After the end, the product will be used for the following 4 months.
  Intervention Group (491 participants): children eating normally, with 2 boxes of Oral Nutritional Supplementation (180ml each) as a snack meal. The product provides 9,5% milk powder, milk fat and 26 micronutrients and provides FOS, HMO, DHA, and Taurine within 4 months of use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): (n=490): children eating normally (not using Oral Nutritional Supplementation) during 4 months of intervention. After the end, the product will be used for the following 4 months.
- Intervention group (Experimental): (n=491): Children eating normally, with 2 boxes of Oral Nutritional Supplementation (180 ml x 2 times/day) as a snack meal.
  The product will be provided for subjects at school 7 days per week (From Monday to Sunday) and at home or school. Children use Oral Nutritional Supplementation twice per day, the first time at 9 am, and the second at 3 pm.
  Interventions: Dietary Supplement: Dielac Grow Plus

INTERVENTIONS:
Dietary Supplement: Dielac Grow Plus — Dialac Grow Plus is an Oral Nutritional Supplementation made by Vietnam Dairy Products Joint Stock Company - Vinamilk.
  Condition: Liquid
  Color: White
  Date of use: 8 months from the manufactured date.
  Preserve: Store in a clean, dry place, and avoid direct sunlight.
  Arms: Intervention group

SUMMARY:
Evaluating the effect of using Oral Nutritional Supplementation toward nutrition status, digestive disorders, upper respiratory disorders, and picky eating in children aged 24 - 59 months.

DETAILED DESCRIPTION:
Evaluating the effect of using Oral Nutritional Supplementation toward improving the nutritional status (anthropometric index, the prevalence of malnutrition) in children aged 24 - 59 months after four months of using the nutritional product.

Evaluating the effect of using Oral Nutritional Supplementation for digestive disorders (diarrhea and constipation), upper respiratory infection and picky eating in children aged 24 - 59 months.

The research involves a randomized controlled clinical trial (RCT), expected from 2023 to 2024 with 1000 children aged 24-59 months. The study will be conducted at schools and homes: 1000 children divided into 2 groups. One group will use the product for 4 months ( with the amount of use: twice per day, 180ml each time). The product will be distributed to the students through the schools. Monitoring will be performed carefully by the commune and district Health Department and the Centers for Disease Control and Prevention weekly. The study aims to evaluate the effect of nutritional products toward nutritional status ( anthropometric index, the prevalence of micronutrients), digestive disorders, and picky eating in children aged 24-59 months.

The nutritional product produces a high amount of energy that provides ≥ 380 kcal/360 ml; 2 bottles equal to 180ml x 2 times/day will provide 28-37,3% energy requirement for children aged 2-4 years old. The product includes fat composition which provides 38-44% energy requirement including 1899 mg medium chain triglyceride (MCT), α Linolenic Acid, Linoleic Acid and 26 types of micronutrients and minerals including some essential micronutrients such as Calcium 110- 130% recommended nutrition needs (RNNs), Iron 58-59,3% RNNs, Vitamin A 91-110% RNNs, Zinc 25-28,9% RNNs, Vitamin D3 54% RNNs, Selen 66-77,6% RNNs, Vitamin K1 27-31,7% RNNs, Folic Acid 72-108% RNNs. Including other compositions such as 2'FL HMO (74 mg), Choline (79mg), Taurine (31,2mg)

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 24 and 59 months old live in 6 selected communes in Yen Bai province.
* The family volunteered for the child to participate in the study
* Z-score height for age <-1 and Z-score weight for height <1
* Participated in the screening and met the selection criteria

Exclusion Criteria:

* Lactose intolerance
* Intellectual disability or suffering from acute and chronic infectious diseases.
* Z-score height for age, Z-score weight for height and Z-score weight for age <-4
* Planing to move out of the selected trials areas in next 6 months

Ages: 24 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 981 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change of anthropometric indicators | After 4 months of intervention
  Children in the intervention group will improve more with the anthropometric indicators (weight, height) than children in the control group.
  This includes weight and height. Weight is measured in kg with one decimal value by the Body composition analyzer called the TANITA scale. Children wear light clothes while measuring. A wooden stadiometer measures height by precisely 0.1cm.
Change of digestive conditions | After 4 months of intervention
  Children in the intervention group will improve more with digestive conditions includes diarrhea, constipation, respiratory infection and picky eating than children in the control group
Change in micronutrients status | After 4 months of intervention
  Children in the intervention group will improve more with the micronutrient status, including the Hb and serum zinc concentrations in blood, than children in the control group.

SECONDARY OUTCOMES:
Change of weight for age Z-score | After 4 months of intervention
  Change of average weight for age Z Score and the difference between before intervention and after the intervention.
  Weight is measured in kg with one decimal value by the Body composition analyzer TANITA scale. The scale is checked and adjusted before use. Children wear light clothing, remove shoes and sandals, and sit or lie balanced, at the center of the scale. As soon as the balance is stable, read and write the result in kg and an odd number after the comma.
  Age of the child is calculated by subtracting the date of birth from the census date and classified according to WHO (World Health Organization) , 2006
Change of weight for height Z-score | After 4 months of intervention
  Change of average weight for height Z Score and the difference between before intervention and after the intervention.
  Weight is measured in kg with one decimal value by the Body composition analyzer TANITA scale. The scale is checked and adjusted before use. Children wear light clothing, remove shoes and sandals, and sit or lie balanced, at the center of the scale. As soon as the balance is stable, read and write the result in kg and an odd number after the comma.
  A wooden stadiometer measures height by precisely 0.1cm. Children stand up straight, their eyes look straight, and the top of their head touches the wooden shelf fixed at a 0 cm position. The child's whole body ensures that 9 points touch the surface of the ruler: occipital, shoulder blade, buttocks, calf, and heel. The result is recorded in centimeter and an odd number after the comma.
Change of height for age Z-score | After 4 months of intervention
  Change of average height for age Z Score and the difference between before intervention and after the intervention.
  A wooden stadiometer measures height by precisely 0.1cm. Children stand up straight, their eyes look straight, and the top of their head touches the wooden shelf fixed at a 0 cm position. The child's whole body ensures that 9 points touch the surface of the ruler: occipital, shoulder blade, buttocks, calf, and heel. The result is recorded in centimeters and an odd number after the comma.
  Age of the child is calculated by subtracting the date of birth from the census date, and classified according to WHO, 2006
Changes in the percentage of children have anorexia, upper respiratory infections or gastrointestinal diseases | After 4 months of intervention
  Changes in the percentage of anorexia, the percentage of gastrointestinal diseases (diarrhea, constipation), and anorexia above after intervention. The changes in digestive disorders would demonstrate in children defecating activities

OTHER OUTCOMES:
Assessment of Caregivers' Perceptions on the Safety and Effectiveness of the Product in Yen Bai | After 4 months of intervention
  Changes in the percentage of anorexia, the percentage of gastrointestinal diseases (diarrhea, constipation), and anorexia above after intervention. The changes in digestive disorders would demonstrate in children defecating activities

CONTACTS AND LOCATIONS:
Overall Officials: Division of Planning National Institute of Nutrition, Principal Investigator — National Institute of Nutrition, Vietnam
Locations (1):
- Yen Bai Province Obstetrics and Children's Hospital, Yên Bái, Vietnam